CLINICAL TRIAL: NCT01311869
Title: Green Tea Extract: a Non-Surgical Alternative for Treatment of Uterine Fibroids
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB Decision
Sponsor: Meharry Medical College (Other)
Responsible Party: Principal Investigator, Ayman Al-Hendy, Principal Investigator, Meharry Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Green Tea Study
Record Dates: First submitted 2011-03-07; First posted 2011-03-10 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Leiomyoma
MeSH Terms: conditions — Leiomyoma | interventions — epigallocatechin gallate; Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGCG ( Green Tea extract) (Active Comparator): 40 subjects will receive 800 mg EGCG orally per day for 6 months versus 40 subjects will receive Brown Rice pill for 6 months
  Interventions: Dietary Supplement: EGCG ( Green Tea extract); Dietary Supplement: Brown rice pills
- Brown Rice pills (Placebo Comparator): 40 subjects will receive 800 mg brown rice pills orally per day for 6 months versus 40 subjects will receive EGCG capsule for 6 months
  Interventions: Dietary Supplement: EGCG ( Green Tea extract); Dietary Supplement: Brown rice pills

INTERVENTIONS:
Dietary Supplement: EGCG ( Green Tea extract) — A randomized double-blind placebo-controlled clinical trial will be conducted with 80 women of reproductive age,the 80 women will be allocated into two groups, 40 each. Each group will be given one of two interventions: The first is 2 capsules of (EGCG which is green tea extract, taken orally with food on daily basis for 6 months, each capsule contain 326.25 mg decaffeinated EGCG,The second group will receive matched (color, taste and texture) placebo for a period of 6 months.
Dietary Supplement: Brown rice pills — 40 subjects will receive 800 mg EGCG orally daily for 6 months, the other 40 subject will receive brown rice pills for the same duration.

SUMMARY:
Uterine Leiomyomata, also known as uterine fibroids, are non-cancer tumors found in the wall of the uterus or womb. Uterine fibroids are the common cause of surgery (removal of the uterus). African American women are 3-4 times more likely to have uterine fibroids. Currently there is no effective long-term medical treatment for fibroids. Hormones have been used for short-term therapy, but they are not used long-term because of the risk of side effects. When women stop receiving the hormone therapy often fibroids return. Surgery is the common treatment for women who are suffering from abnormal symptoms caused by fibroids. Hysterectomy is an effective treatment, however women cannot have children after removal of the uterus.

Epigallocatechin Gallate (EGCG) is one of the main natural chemicals found in green tea.. Research the investigators have done in the laboratory and in animals leads them to believe EGCG may decrease the growth of fibroids.

This study is intended to determine whether EGCG will cause fibroid tumors to shrink and reduce fibroid related symptoms such as abnormal vaginal bleeding and pelvic discomfort.

DETAILED DESCRIPTION:
* Uterine leiomyoma (also known as fibroids) are benign estrogen-dependent tumors of the uterine wall. Uterine fibroids are the most common tumors of the female reproductive tract, occurring in 20-70% of premenopausal women in the reproductive age women and cause multiple clinical complications such as acute and chronic pelvic pain as well as excessive vaginal bleeding and iron deficiency anemia, moreover they are considered as the leading indication for hysterectomy in reproductive age African American (AA) women. The impact of these serious clinical complications on women's health is tremendous. African American women are particularly affected as the prevalence of uterine fibroids is about 4 times higher in that ethnic group compared to Caucasians. Being a major health disparity issue, uterine fibroids appear to further diminish the quality of life for AA women who also suffer from higher incidence of chronic diseases such as diabetes, heart disease, obesity, and cancer. Currently there is no effective long-term medicinal treatment for this common disease. GnRH analogues are effective short medical therapy option. However, they are not approved for long-term (more than 3 months) because of the risk of irreversible bone loss and osteoporosis and other major side effects. When these medications are discontinued, the fibroids return to their original size with symptoms recurring, that is why they are FDA approved in uterine fibroids only as preoperative adjuvant to improve the fibroid-related iron-deficiency anemia. Surgery, usually in the form of hysterectomy, is the traditional treatment of women with symptomatic uterine fibroids. Clearly hysterectomy is an effective treatment but it precludes future fertility. This creates a major dilemma for women with symptomatic uterine fibroids who have not completed their families or have not even started a family. Problems with fibroids must be viewed as a public health concern as well as a major health disparity issue. The general public in relation to this problem must be concerned about the: (1) The decrease in the quality of life of women who are affected, and hence the well-being of the whole family; (2) Interference with inter-family dynamics and relationships. Decrease in productivity in the workforce/job performance. Increase in cost of health care caused by the more than 600,000 hysterectomies/Y in USA alone.
* Green Tea Extract

This work will evaluate the utility of EGCG, green tea extract, which is a common nutritional supplement, in symptomatic relief of this common women's health problem. Considering the wide acceptability of nutritional supplements especially among African American women, the ethnic group most affected by uterine fibroids, this project can potentially provide an effective and inexpensive non-surgical alternative for management of uterine fibroids. Green tea is a common agent used by women for multiple purposes. Epigallocatechin gallate (EGCG) is the major catechin (about 80%) of green tea. EGCG exhibit several useful biological effects including anti-inflammatory, anti-proliferative as well as anti-oxidant effects. A study conducted by the United States Department of Agriculture reported that green tea has potent anti-cancer effects against a wide range of human cancer cells. Green tea's polyphenols, most notably EGCG, are considered responsible for those positive effects. Green tea polyphenols have also been shown to inhibit key pathways of tumor growth.

* Prior Human Experience with EGCG Several human clinical studies used EGCG for extended periods of time in which EGCG was very well tolerated with virtually no reportable side effects. Wolfarm and colleagues used oral EGCG 300 mg/day in cardiac patients and reported improved endothelial function and increased brachial artery flow-mediated dilation that paralleled changes in EGCG plasma concentration. reported on the consumption of 500-1000 mg/day of oral EGCG for 3 months which resulted in marked decrease in several anti-oxidative biomarkers compared to placebo. Numerous studies have described favorable effects of EGCG when used in overweight and obese individuals for extended durations. Chow et.al. reported on human use of EGCG with 30 healthy volunteers randomly assigned to one of the following doses of Polyphenon E (a decaffeinated green tea catechin mixture): 400, 800, or 1200 mg/day (10 subjects per dose group). Only transient mild nausea was noted in 3% of the study participants and was seen only at the highest study agent dose (1200 mg EGCG/day) and in the fasting condition. Doses of 800mg were well tolerated with no reported side effects. Grapes also contain polyphenols and catechins such as EGCG. EGCG is the most powerful of these catechins that accounts for the favorable health effects from the use of grapes extracts. Grapes polyphenols have been shown to inhibit key pathways of tumor growth. Grapes EGCG appear to block each stage of tumor-genesis by modulating signaling pathways involved in cell proliferation, transformation, inflammation, and oxidative stress, which are clearly involved in pathogenesis of various tumors including uterine fibroids. Freeze-dried table grapes powder has been used recently for several months in pre-and post-menopausal women at doses of up to 36 gm/day. This dose corresponds to about 800mg EGCG/day. This treatment was very well tolerated with no reported side effects. This suggests that such supplement can be successfully administered to women as part of life or diet modification programs.
* Preclinical Data Recent studies from our group demonstrated the ability of EGCG to control the proliferation and to induce apoptosis in human leiomyomata cells in vitro and in animal models. Our preclinical data in fibroid animal models demonstrates that EGCG at a dose of 1.25mg/Kg/day added to drinking water was able to induce a highly significant (up to 80%) shrinkage of fibroid lesions compared to untreated controls. The treatment was well tolerated with no detected side effects. Such daily doses of EGCG have been administered safely to human subjects in prior clinical trials. This effect is partially attributed to potent inhibitory effect of EGCG on Catechol-O-methyl transferase (COMT), an enzyme that we have recently linked to pathogenesis of uterine fibroids. In this proposal we aim to evaluate the efficacy of Epigallocatechin gallate (EGCG) in reducing the size of uterine fibroids and improving quality of life in women with symptomatic uterine fibroids, as well as assess its safety profile.
* We have recently demonstrated elevated levels of expression of catechol-O-methyl transferase (COMT) in uterine fibroids compared to adjacent normal myometrium, and described its important role in fibroid pathogenesis.
* Interestingly, recent reports demonstrated that EGCG has potent anti-COMT activity. These reports have shown that green tea extract intake is associated with weight loss due to diet-induced thermo-genesis. This effect is generally attributed to EGCG. This catechin is known to be capable of inhibiting COMT, which is the enzyme that degrades nor-epinephrine, thus stimulating thermo-genesis. The inhibition of COMT by EGCG was uncompetitive with respect to S-adenosylmethionine (SAM) suggesting that there is no direct interaction between EGCG and the SAM-binding site on the COMT, yet there was clear inhibition of COMT activity with increasing EGCG concentration. Additionally, the Vmax values for methylation were decreased. Our preliminary data also showed that EGCG inhibited COMT gene expression in a dose-dependent manner in human leiomyomata cells.
* Our hypothesis is that the use of the "EGCG" as a nutritional supplement will decrease the size of uterine fibroids and improve fibroids-related clinical symptoms in women resulting in a significant improvement in their quality of life.
* This work will evaluate the utility of a common nutritional supplement in symptomatic relief of a very common women's health problem. Considering the availability, lower cost, as well as the wide acceptability of nutritional supplements, this project can potentially provide an inexpensive non-surgical alternative for management of uterine fibroids which would have a major impact on health of women from all ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* Female; Age: 18Y or older.
* Pre-menopausal.
* FSH level is less than 10 mIU/L.
* Have at least moderate uterine fibroid-related symptoms (score of 24 or higher according to UFS-QOL questionnaire.
* Have a total uterine volume greater than or equal to 160 cc by ultrasound measurement and at least one fibroid that is ≥ 2.5cm in diameter.
* Agree to use a double-barrier method (condoms, diaphragms) or other effective non-hormonal methods of contraception (abstinence, sterilization) throughout participation in the study to prevent pregnancy.
* Agree to report any pregnancy to the research staff immediately.
* Willing and able to give informed consent.
* Willing and able to comply with study requirements.
* Liver function (ALT, AST, Prothrombin time and concentration)to be≤ 1.5 times the upper limit of normal

Exclusion Criteria:

* Current or planned pregnancy during the study period.
* Menopausal, as indicated by elevated follicle stimulating hormone (FSH) serum level.
* Currently breast-feeding.
* Untreated abnormal pap smear.
* Presence of conditions other than fibroids contributing to pelvic pain and/or bleeding;
* Hemoglobin < 8.0 mg/dl.
* Presence of adnexal masses or tenderness indicating the need for further evaluation or surgery.
* Grade III or IV hydronephrosis by ultrasound.
* Mental health disorder.
* Active substance abuse or dependence.
* Current or recent (within the past 3 months) use of the following medications: Oral or systemic corticosteroids, Hormones (estrogen, progestins, oral contraceptives), Danazol, anticoagulants, Herbal or botanical supplements with possible hormonal or EGCG effects. Use within the past six months of the gonadotropin releasing hormones (GnRH) analogs or Depo-Provera,
* Current or planned use during the study of any of the following medications/or products: ketoconazole, itraconazole, erythromycin, grapefruit juice, rifampin, St John's Wort, phenytoin, phenobarbital, or carbamazepine.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
fibroid size | 6 months

SECONDARY OUTCOMES:
Quality of life | Every month for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Al-Hendy, MD, PhD, Principal Investigator — Meharry Medical College
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Johnson JJ, Siblini H, Al-Hendy A, Segars JH, Gonzalez F, Taylor HS, Singh B, Carson SA, Christman GM, Huang H, Dangi B, Zhang H. Evaluating the Effect of Epigallocatechin Gallate (EGCG) in Reducing Folate Levels in Reproductive Aged Women by MTHFR and DHFR Genotype in Combination With Letrozole or Clomiphene. Clin Transl Sci. 2025 Mar;18(3):e70189. doi: 10.1111/cts.70189. PMID 40077973